CLINICAL TRIAL: NCT01076842
Title: The Effect of Detemir Compared to Exenatide and/or the Combination of Detemir and Exenatide on Glycemic Control and Weight in Patients With Type 2 Diabetes Mellitus Who Have Failed Oral Hypoglycemic Agents
Brief Title: Efficacy Evaluation of Different Medication Combination in Type 2 Diabetes Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Collaborators: BodyMedia (Unknown)
Responsible Party: Col. Robert A. Vigersky, MD MC, WRAMC- Diabetes Institute
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-13028
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Type 2
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Detemir; Exenatide; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A Levemir (Active Comparator): Levemir once daily, force titrated to reach a fasting plasma glucose of 100 mg/dl
  Interventions: Drug: Insulin-Levemir; Device: SenseWear Pro3® armband; Device: DexCom CGM
- B Exenatide (Active Comparator): Exenatide twice daily, started at a dose of 5 mcg b.i.d. and increased to 10 mcg b.i.d. after 2 weeks if the fasting plasma glucose of 100 mg/dl is not reached. Exenatide will be administered immediately before breakfast and dinner meals. No further increase in the dose of exenatide will take place. For those who are unable to tolerate exenatide at a 10 mcg b.i.d. dose, it will be reduced to 5 mcg b.i.d. and continued until week 12.
  Interventions: Drug: Exenatide-Bayetta; Device: SenseWear Pro3® armband; Device: DexCom CGM
- C Levemir+Exenatide (Active Comparator): Patients from either Group A or Group B who have not reached the goal A1C of 6.5% will be assigned to this Group. They will receive the drug assigned to the other group in addition to the one they were originally assigned.
  Interventions: Drug: Insulin-Levemir and Exenatide-Bayetta; Device: SenseWear Pro3® armband; Device: DexCom CGM

INTERVENTIONS:
Drug: Insulin-Levemir — Levemir once daily, force titrated to reach a fasting plasma glucose of 100 mg/dl
  Other Names: Levemir
  Arms: A Levemir
Drug: Exenatide-Bayetta — Exenatide twice daily, started at a dose of 5 mcg b.i.d. and increased to 10 mcg b.i.d. after 2 weeks if the fasting plasma glucose of 100 mg/dl is not reached. Exenatide will be administered immediately before breakfast and dinner meals. No further increase in the dose of exenatide will take place. For those who are unable to tolerate exenatide at a 10 mcg b.i.d. dose, it will be reduced to 5 mcg b.i.d. and continued until week 12.
  Other Names: Exenatide
  Arms: B Exenatide
Drug: Insulin-Levemir and Exenatide-Bayetta — Patients from either Group A or Group B who have not reached the goal A1C of 6.5% will be assigned to this Group. They will receive the drug assigned to the other group in addition to the one they were originally assigned.
  Other Names: Levemir+Exenatide
  Arms: C Levemir+Exenatide
Device: SenseWear Pro3® armband — For one-week prior to beginning the assigned medication and for one week , week 11 and week 23, the patients will wear the SenseWear Pro3® armband for collection of ancillary physiologic data
  Other Names: armband
Device: DexCom CGM — For one-week prior to beginning the assigned medication and for one week , week 11 and week 23, the patients will wear the DexCom CGM for collection of continuous blood glucose concentrations.
  Other Names: continuous glucose monitoring

SUMMARY:
The purpose of this study is to compare the effectiveness of two different kinds of diabetes medications, insulin detemir (Levemir) and exenatide (Byetta), in improving blood sugar levels with little or no weight gain in patients with type 2 diabetes who are not well controlled on two or more oral (by mouth) diabetes medications. Both medications are given by injection with a very small needle just below the surface of your skin (called subcutaneous injection). The medication that you inject will be in addition to your oral medications.

DETAILED DESCRIPTION:
Finding a safe and effective method of improving blood glucose (BG) control without weight gain is one of the major goals of diabetes research. Previous research studies have shown that Levemir and Byetta are safe and effective medications in the treatment of type 2 diabetes. Both drugs have been approved by the U.S. Food and Drug Administration (FDA) for the treatment of type 2 diabetes. The use of Levemir and Byetta in combination in this study, is investigational, meaning it is not approved by the FDA for this use. However, the FDA has allowed the use of Levemir and Byetta in combination in this study of safety and effectiveness in improving blood sugar levels with little or no weight gain in people with type 2 diabetes.

Levemir is a long acting insulin that is usually taken once a day at bedtime and can last for up to 24 hours. Unlike most insulins that lower blood glucose levels, but cause weight gain, clinical research trials suggest that Levemir may lower blood glucose levels without causing weight gain and may even result in weight loss.

Byetta is not insulin, but improves blood glucose control by mimicking the action of hormones in the gastrointestinal tract called incretins. The incretin hormones trigger the release of insulin from the pancreas and allow insulin to work more effectively in the body. Byetta also delays the movement of food from the stomach into the small intestine. As a result, people taking Byetta may feel "full" faster and longer, so they eat less. The most common side effect with Byetta is mild to moderate nausea, which improves with time in most people. Clinical research trials that have studied the effects of Byetta have shown that, in addition to lowering blood glucose levels, the use of Byetta resulted in weight loss.

There have been no previous studies that have compared Levemir to Byetta in patients who have failed to achieve blood glucose goals with two or three oral diabetes medications.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Type 2 DM for over six months
2. A history of inadequate glycemic control (A1c > 7.5% but < 10%) despite treatment with 2 or more oral hypoglycemic agents
3. 18 years of age or older
4. Stable medical status (e.g., no myocardial infarction, stroke, major surgery, or major mental illness during the previous 6 months)
5. Naïve to insulin (no insulin for more than 14 days during the previous 6 months and none within 60 days of beginning the study)
6. On at least ½ maximum or the greatest tolerable dose of their oral agents according to the label for at least 3 months
7. BMI < 40 kg/m2
8. Willing to perform at least four finger stick blood glucose measurements each day

Exclusion Criteria:

1. A diagnosis of Type 2 DM for less than six months
2. An A1c of < 7.5% or > 10%
3. Pregnancy as determined by a serum ß HCG.
4. An unstable medical status
5. Taking glucocorticoids, amphetamines, anabolic, or weight-reducing agents during the course of the study
6. Inability to read and write English
7. Someone who is not likely to return for the follow-up because they or their sponsor is likely to have a permanent change of station or termination of service before completion of the protocol
8. Unwilling to perform four finger stick blood glucose measurements each day
9. Previous history of use of exenatide

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the improvement in A1C goal measured in mean reduction in A1c levels over 24 weeks. | 1 month

SECONDARY OUTCOMES:
Hypoglycemia weight waist-hip ratio frequency of hypoglycemia weight FBGL lipid levels CBC CMP biometric parameters of activity heat flux galvanic skin response heart rate level of physical activity and energy expenditure | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Vigersky, MD, Principal Investigator — WRAMC- Diabetes Institute
Locations (2):
- United States (2):
  - MedStar Research Institute, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia